CLINICAL TRIAL: NCT05951387
Title: Comparative Study of Hemodynamic Changes and Sedation Effect of Dexmedetomidine Versus Dexmedetomidine with Ketamine in Mechanically Ventilated ARDS Patients, Randomized Clinical Trial
Brief Title: Dexmedetomidine Versus Dexmedetomidine with Ketamine in Mechanically Ventilated ARDS Patients
Acronym: ARDS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Marwa Elsayed Elnaggar, Assistant professor of chest diseases, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RC 37-5-2023
Record Dates: First submitted 2023-06-14; First posted 2023-07-19 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2023-07

CONDITIONS: Haemodynamic Instability
Keywords: ARDS; Dexmedetomidine; ketamine
MeSH Terms: interventions — Dexmedetomidine; Ketamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- dexmedetomidine plus ketamine (Active Comparator): starting intravenous infusion dose of dexmedetomidine 0.5 µg/kg/h mixed with ketamine 0.5 mg/kg/h to 30 mechanically ventilated ARDS patient
  Interventions: Drug: dexmedetomidine plus ketamine
- high dose dexmedetomidine (Active Comparator): dexmedetomidine at 0.5 µg/kg/h intravenous infusion only to be titrated to achieve full sedation to 30 mechanically ventilated ARDS patient
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: dexmedetomidine plus ketamine — titrating the dose of dexmedetomidine mixed with ketamine (staring dose 0.5ug/kg/hr, 0.5mg/kg/hr respectively)to achieve full sedation
  Other Names: Group A
  Arms: dexmedetomidine plus ketamine
Drug: Dexmedetomidine — starting intravenous infusion with dexmedetomidine starting at dose 0.5ug/kg//hr and titrate the dose to achieve full sedation
  Other Names: Group B
  Arms: high dose dexmedetomidine

SUMMARY:
The goal of this clinical trial study is to compare dexmedetomidine versus the combination of dexmedetomidine with ketamine in hemodynamic changes and sedative effects in ARDS patients who are in need of mechanical ventilation. The main question[s] it aims to answer are:

* [question 1]: Which dose that get the target in sedation, single and combined drugs?
* [question 2]: In which drug group that hemodynamic did not affect Participants will be patients with ARDS that will be divided into two group the first ont will receive dexmedetomidine 0.5 µg/kg/h mixed with ketamine 0.5 mg/kg/h and the second one will receive dexmedetomidine at 0.5 µg/kg/h infusion only. In both the groups, studied drugs will be titrated to achieve target sedation.

DETAILED DESCRIPTION:
This study will include 60 patients with ARDS who will be admitted to the intensive care unit (ICU) and chest ICU of Banha university hospitals during the period between June 2023 and June 2024.

ARDS will be diagnosed based on the presence of new or worsening symptoms within one week of a known clinical insult; bilateral opacities on anteroposterior chest X-ray that are not due to effusions, nodules or lobar or lung collapse; and hypoxemia, defined as arterial oxygen tension/fraction of inspired oxygen (Pao2/FiO2) < 300 mm Hg and a minimum positive end-expiratory pressure ≥ 5 cm H2O, that is not explained by heart failure or fluid overload.

Patients were divided randomly into two groups. Group A (n = 30); received with starting dose of dexmedetomidine 0.5 µg/kg/h mixed with ketamine 0.5 mg/kg/h and Group B (n = 30); received dexmedetomidine at 0.5 µg/kg/h infusion only. In both the groups, studied drugs will be titrated to achieve target sedation.

All patients will be subjected to the following:

1. Thorough history taking and clinical examination
2. Calculation of acute physiology and chronic health evaluation (APACHE) score at time of ICU admission
3. Sedation score calculation using the Richmond Agitation-Sedation Scale (RASS)
4. ECG, blood pressure monitoring
5. Measurement of plasma C-reactive protein (CRP) level before and after initiation of sedation.
6. Measurement of oxygenation status (Pao2/Fio2) before and at 24, 48, 72, and 120 h after the administration of the sedatives
7. Any adverse effects related to sedation or intubation will be recoded

All data will be tabulated and statistically analyzed

ELIGIBILITY:
Inclusion Criteria:

* patients with ARDS with the following:

  * Those whose duration of endotracheal intubation was > 120 h
  * those whose ages were 18- 70 years old
  * those with acute physiology and chronic health evaluation (APACHE) II scores > 12 points.

Exclusion Criteria:

* patients with a history of allergy to ketamine or dexmedetomidine
* Pregnant women,
* patients in the early stage of recovery,
* patients with unstable hemodynamics, bradycardia, sinus arrest, or other cardiac arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
oxygenation parameter | 24-27 hours
  change of PaO2/FiO2
positive end expiratory pressure (PEEP) | 24-27 hours
  change of PEEP parameter that need to maintain oxygen saturation above 88%

SECONDARY OUTCOMES:
serum level of C-reactive protein (CRP) | 24-72 hours
  change of serum level of CRP (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Elnaggar, MD, Study Director — Benha University, Faculty of medicine
Locations (1):
- Benha university, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No